CLINICAL TRIAL: NCT05631613
Title: Transarterial Chemoembolization With Lipiodol-Idarubicin Emulsion Based On a Specific Ratio for Hepatocellular Carcinoma:a Prospective, Observational Study
Brief Title: Lipiodol-TACE With Idarubicin Based On a Specific Emulsion Ratio for Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, President, Zhongda Hospital
Other Study IDs: Idarubicin-cTACE
Record Dates: First submitted 2022-08-15; First posted 2022-11-30 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Transarterial chemoembolization; Idarubicin; Lipiodol emulsion; prospective study
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Water for Injection -Idarubicin -Lipiodol: Idarubicin is first dissolved in water for injection to make a solvent of
  1mg/ml, which is then mixed with lipiodol to make an emulsion with a ratio of 1:2. Lipiodol-idarubicin emulsion is slowly injected, followed by embolization with embolic agents.
  Interventions: Procedure: cTACE(conventional transarterial chemoembolization)
- Nonionic Contrast Agent -Idarubicin -Lipiodol: Idarubicin is first dissolved in nonionic contrast agent to make a solvent of
  1mg/ml, which is then mixed with lipiodol to make an emulsion with a ratio of 1:2. Lipiodol-idarubicin emulsion is slowly injected, followed by embolization with embolic agents.
  Interventions: Procedure: cTACE(conventional transarterial chemoembolization)

INTERVENTIONS:
Procedure: cTACE(conventional transarterial chemoembolization) — transarterial chemoembolization with lipiodol-idarubicin emulsion

SUMMARY:
The purpose of this observational study is to evaluate properties of lipiodol-idarubicin emulsion mixed with the best regimen obtained in vitro study, including stability, viscosity，visibility under X-ray and deposition, in order to maximize the efficacy of idarubicin-cTACE for HCC.

DETAILED DESCRIPTION:
Idarubicin is a DNA topoisomerase II inhibitor that promotes DNA strand breakage, trapping cells in the G2 phase of the cell cycle and inducing DNA cleavage and cell apoptosis. Preclinical studies have shown that idarubicin has higher antitumor activity than epirubicin, especially against SUN-449 human hepatoma cells.

In recent years, foreign scholars have conducted a series of explorations in the treatment of hepatocellular carcinoma with lipiodol-idarubicin emulsion, and have obtained positive results.

However, in China, idarbicin has just been applied to TACE.Many interventional physicians are accustomed to directly use contrast agents to dissolve anthracyclines in order to improve tracer performance of chemotherapeutic agent-lipiodol emulsion under X-ray and reduce intraoperative reflux and misembolization. Meanwhile, due to the high density of the nonionic contrast media, the lipiodol emulsion can be deposited in the lesion for a long time. The Clinical Practice Guidelines for transcatheter arterial chemoembolization (TACE) Treatment of hepatocellular carcinoma in China (2021 edition) also recommended to prepare the chemotherapeutic drug-lipiodol emulsion according to the standard of " dissolving drug in nonionic contrast agent then mixed with lipiodol to make an emulsion with a ratio of 1:2".

At present, there is a lack of detailed objective data on the complete physical properties of the lipiodol-idarubicin emulsion, and some physicians and centers even make the emulsion based only on their habits and preferences.These all may affect the physical properties of the lipiodol emulsion, including intraoperative stability and viscosity of the emulsion, then eventually affect the operation of surgeon and the release behavior of chemotherapeutic drugs, and ultimately influence the efficacy of TACE.Therefore, the purpose of this prospective, observational study is to evaluate properties of lipiodol-idarubicin emulsion mixed with the best regimen obtained in vitro study, including stability, viscosity，visibility under X-ray and deposition, in order to maximize the efficacy of idarubicin-cTACE for HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of HCC according to histopathology or CNLC guidelines (2022 Edition);
2. One of the following cases:

1）CNLC stage IIb-IIIa, part of stage IIIb, and CNLC stage Ib and IIa patient who is unable or unwilling to receive surgical treatment due to other reasons (such as advanced age, severe liver cirrhosis, etc.); 2).Child-Pugh class A or B; 3).ECOG PS of 0 - 2; 4)The main portal vein has not been completely obstructed, with abundant collateral vessels, or restore the blood flow by portal vein stent placement 3.At least one measurable lesion (enable to assess lipiodol deposition); 4.Be willing to participate in this study.

Exclusion Criteria:

1. Non-HCC patients treated with TACE
2. Incomplete clinical and imaging data
3. Poor image quality or other difficulties in assessing intratumoral lipiodol deposition, including:

1) A large amount of lipiodol was deposited around the lesion 2) Diffuse tumor distribution 3) Intratumoral lipiodol deposition from previous TACE 4) Metal artifacts from previous operations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated by lipiodol TACE with idarubicin for HCC
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Deposition of of lipiodol-idarubicin emulsion | intraoperative and up to 7 days
  1. Assessed by two or more senior radiologists as described in previous works: Excellent：>90%；Good：50%-90%；Poor：<50% 2.3D quantitative assessments of intratumoral lipiodol-emusion using the software 3d-slicer： V1=Volume of tumor (cm3) V2=volume of lipiodol deposition (cm3) Degree of iodized oil uptake:Intratumoral lipiodol retention(%)=V1/V2

SECONDARY OUTCOMES:
Stability of lipiodol-idarubicin emulsion | intraoperative
  Observe and assess the separation of emulsion（when it occures, record the percentage of aqueous phase, the persisting emulsion and the oily phase）
Viscosity of lipiodol-idarubicin emulsion | intraoperative
  Observe the tube-adhesion of emulsion.The subjective perception of injection is evaluated by questionnaire.
Visibility of lipiodol-idarubicin emulsion under X-ray: image quality | intraoperative and up to 7 days
  Assessed by two or more senior radiologists according to Subjective Relative Evaluation of Images.

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Dong Zhu, MD, Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Mak LY, Wong DK, Pollicino T, Raimondo G, Hollinger FB, Yuen MF. Occult hepatitis B infection and hepatocellular carcinoma: Epidemiology, virology, hepatocarcinogenesis and clinical significance. J Hepatol. 2020 Oct;73(4):952-964. doi: 10.1016/j.jhep.2020.05.042. Epub 2020 Jun 3. PMID 32504662
- [Background] Allemani C, Matsuda T, Di Carlo V, Harewood R, Matz M, Niksic M, Bonaventure A, Valkov M, Johnson CJ, Esteve J, Ogunbiyi OJ, Azevedo E Silva G, Chen WQ, Eser S, Engholm G, Stiller CA, Monnereau A, Woods RR, Visser O, Lim GH, Aitken J, Weir HK, Coleman MP; CONCORD Working Group. Global surveillance of trends in cancer survival 2000-14 (CONCORD-3): analysis of individual records for 37 513 025 patients diagnosed with one of 18 cancers from 322 population-based registries in 71 countries. Lancet. 2018 Mar 17;391(10125):1023-1075. doi: 10.1016/S0140-6736(17)33326-3. Epub 2018 Jan 31. PMID 29395269
- [Background] Reig M, Forner A, Rimola J, Ferrer-Fabrega J, Burrel M, Garcia-Criado A, Kelley RK, Galle PR, Mazzaferro V, Salem R, Sangro B, Singal AG, Vogel A, Fuster J, Ayuso C, Bruix J. BCLC strategy for prognosis prediction and treatment recommendation: The 2022 update. J Hepatol. 2022 Mar;76(3):681-693. doi: 10.1016/j.jhep.2021.11.018. Epub 2021 Nov 19. PMID 34801630
- [Background] Lu J, Zhao M, Arai Y, Zhong BY, Zhu HD, Qi XL, de Baere T, Pua U, Yoon HK, Madoff DC, Teng GJ; International Society of Multidisciplinary Interventional Oncology (ISMIO). Clinical practice of transarterial chemoembolization for hepatocellular carcinoma: consensus statement from an international expert panel of International Society of Multidisciplinary Interventional Oncology (ISMIO). Hepatobiliary Surg Nutr. 2021 Oct;10(5):661-671. doi: 10.21037/hbsn-21-260. PMID 34760969
- [Background] Chen C, Lu L, Yan S, Yi H, Yao H, Wu D, He G, Tao X, Deng X. Autophagy and doxorubicin resistance in cancer. Anticancer Drugs. 2018 Jan;29(1):1-9. doi: 10.1097/CAD.0000000000000572. PMID 29099416
- [Background] Zhong S, Li C, Han X, Li X, Yang YG, Wang H. Idarubicin Stimulates Cell Cycle- and TET2-Dependent Oxidation of DNA 5-Methylcytosine in Cancer Cells. Chem Res Toxicol. 2019 May 20;32(5):861-868. doi: 10.1021/acs.chemrestox.9b00012. Epub 2019 Mar 11. PMID 30816036
- [Background] Armenian S, Bhatia S. Predicting and Preventing Anthracycline-Related Cardiotoxicity. Am Soc Clin Oncol Educ Book. 2018 May 23;38:3-12. doi: 10.1200/EDBK_100015. PMID 30231396
- [Background] Feng F, Jiang Q, Jia H, Sun H, Chai Y, Li X, Rong G, Zhang Y, Li Z. Which is the best combination of TACE and Sorafenib for advanced hepatocellular carcinoma treatment? A systematic review and network meta-analysis. Pharmacol Res. 2018 Sep;135:89-101. doi: 10.1016/j.phrs.2018.06.021. Epub 2018 Jun 26. PMID 29959032
- [Background] Mizutani H, Shiga C, Imai M, Ikemura K, Kitamura Y, Ohta K, Miyazawa D, Sakanashi M, Tahira T, Maeda T, Hiraku Y, Kawanishi S. Idarubicin, an Anthracycline, Induces Oxidative DNA Damage in the Presence of Copper (II). Anticancer Res. 2020 Oct;40(10):5399-5404. doi: 10.21873/anticanres.14548. PMID 32988859
- [Background] Boulin M, Guiu S, Chauffert B, Aho S, Cercueil JP, Ghiringhelli F, Krause D, Fagnoni P, Hillon P, Bedenne L, Guiu B. Screening of anticancer drugs for chemoembolization of hepatocellular carcinoma. Anticancer Drugs. 2011 Sep;22(8):741-8. doi: 10.1097/CAD.0b013e328346a0c5. PMID 21487286
- [Background] Boulin M, Schmitt A, Delhom E, Cercueil JP, Wendremaire M, Imbs DC, Fohlen A, Panaro F, Herrero A, Denys A, Guiu B. Improved stability of lipiodol-drug emulsion for transarterial chemoembolisation of hepatocellular carcinoma results in improved pharmacokinetic profile: Proof of concept using idarubicin. Eur Radiol. 2016 Feb;26(2):601-9. doi: 10.1007/s00330-015-3855-4. Epub 2015 Jun 11. PMID 26060065
- [Background] Favelier S, Boulin M, Hamza S, Cercueil JP, Cherblanc V, Lepage C, Hillon P, Chauffert B, Krause D, Guiu B. Lipiodol trans-arterial chemoembolization of hepatocellular carcinoma with idarubicin: first experience. Cardiovasc Intervent Radiol. 2013 Aug;36(4):1039-46. doi: 10.1007/s00270-012-0532-8. Epub 2012 Dec 8. PMID 23224215
- [Background] Tavernier J, Fagnoni P, Chabrot P, Guiu B, Vadot L, Aho S, Boyer L, Abergel A, Hillon P, Sautou V, Boulin M. Comparison of two transarterial chemoembolization strategies for hepatocellular carcinoma. Anticancer Res. 2014 Dec;34(12):7247-53. PMID 25503156
- [Background] Guiu B, Jouve JL, Schmitt A, Minello A, Bonnetain F, Cassinotto C, Piron L, Cercueil JP, Loffroy R, Latournerie M, Wendremaire M, Lepage C, Boulin M. Intra-arterial idarubicin_lipiodol without embolisation in hepatocellular carcinoma: The LIDA-B phase I trial. J Hepatol. 2018 Jun;68(6):1163-1171. doi: 10.1016/j.jhep.2018.01.022. Epub 2018 Feb 8. PMID 29427728
- [Background] Tzeng WS, Wu RH, Chang SC, Chou CK, Lin CY, Chen JJ, Yang SC, Lin CH. Ionic versus nonionic contrast media solvents used with an epirubicin-based agent for transarterial chemoembolization of hepatocellular carcinoma. J Vasc Interv Radiol. 2008 Mar;19(3):342-50. doi: 10.1016/j.jvir.2007.10.021. PMID 18295692
- [Background] Wang Z, Chen R, Duran R, Zhao Y, Yenokyan G, Chapiro J, Schernthaner R, Radaelli A, Lin M, Geschwind JF. Intraprocedural 3D Quantification of Lipiodol Deposition on Cone-Beam CT Predicts Tumor Response After Transarterial Chemoembolization in Patients with Hepatocellular Carcinoma. Cardiovasc Intervent Radiol. 2015 Dec;38(6):1548-56. doi: 10.1007/s00270-015-1129-9. Epub 2015 May 23. PMID 26001366
- [Background] Letzen BS, Malpani R, Miszczuk M, de Ruiter QMB, Petty CW, Rexha I, Nezami N, Laage-Gaupp F, Lin M, Schlachter TR, Chapiro J. Lipiodol as an intra-procedural imaging biomarker for liver tumor response to transarterial chemoembolization: Post-hoc analysis of a prospective clinical trial. Clin Imaging. 2021 Oct;78:194-200. doi: 10.1016/j.clinimag.2021.05.007. Epub 2021 May 18. PMID 34022765